CLINICAL TRIAL: NCT01530425
Title: Development of a Suite of Outcomes Measures Suitable for Use in Low-resource Settings to Compare Pediatric Wheelchairs Within the Framework of the International Classification of Function, Disability and Health
Brief Title: Outcome Measures for Pediatric Wheelchairs in Low-resource Settings
Acronym: Wheels
Status: Terminated | Type: Observational
Why Stopped: sufficient info
Sponsor: Bethany Relief and Rehabilitation International Inc. (Other)
Collaborators: LeTourneau University (Other); Queen's University (Other)
Responsible Party: Sponsor
Other Study IDs: BKK-WRWC
Record Dates: First submitted 2011-06-21; First posted 2012-02-10 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2015-02

CONDITIONS: Shoulder Impingement; Pressure Ulcer
Keywords: pediatric wheelchairs; low-income; comparisons
MeSH Terms: conditions — Shoulder Impingement Syndrome; Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Phase 1 assessments: Regency Wheelchairs and APDK 12-inch wide wheelchairs
- Phase 2 assessments: Hope Haven and APDK 14-16 inch wide wheelchairs
- Phase 3 assessments: Motivation and Whirlwind wheelchairs

SUMMARY:
Two wheelchair types available for children in Kenya are assessed for energy costs, utility, and complications. This study will arrive at a protocol for assessing wheelchairs in low-income settings, and in the process, provide wheelchair makers and providers with specific feedback. It also serves as a means to increase the skills of local health professionals working with the children in this study, while providing them with appropriate wheelchairs to use.

DETAILED DESCRIPTION:
In each of 2011, 2012, and 2013, two different low cost wheelchairs were assessed. User feedback, health professional feedback, and objective measures were employed for these assessments in the real world setting. Participants for each phase were recruited from a Kenyan Primary or Secondary Schools for children with disability.

ELIGIBILITY:
Inclusion Criteria:

* Children who would benefit from available study wheelchairs who are able to provide feedback

Exclusion Criteria:

* Children who are not able to provide feedback on the study wheelchairs

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with disabilities in a primary school in Kenya who would benefit from available study wheelchairs, and who can provide feedback. Assent provided with parental consent.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
physiologic costs (FEW) | within 1 year of wheelchair acquisition for each phase
  energy costs will be measured, feedback will be obtained from children (VAS)

SECONDARY OUTCOMES:
medical complications | within 24 months after wheelchair distribution for each phase
  direct assessment by physician for Musculoskeletal and Skin complications
participation | within 24 months after wheelchair distribution for each phase
  using decriptive data to describe effect of wheelchair use on participation in school and play

CONTACTS AND LOCATIONS:
Overall Officials: Karen Rispin, Principal Investigator — LeTourneau University
Locations (1):
- Kenyan Primary School, Thika, Kenya